CLINICAL TRIAL: NCT01608581
Title: Development and Evaluation of an Adult Burn Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Responsible Party: Principal Investigator, Jennifer Paratz, Research Chair, Burns Trauma Critical Care Research Centre, The University of Queensland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: flaming fool
Record Dates: First submitted 2012-05-22; First posted 2012-05-31 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Burns
Keywords: prevention; burn; adult; health promotion; evaluation; media
MeSH Terms: conditions — Burns | interventions — Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- exposure to multi-media campaign (Experimental): A multimedia campaign highlighting dangers of gasoline and fire was delivered to an intervention region in the state of Queensland
  Interventions: Other: multimedia burn awareness campaign

INTERVENTIONS:
Other: multimedia burn awareness campaign — Television commercials x4 delivered 86 times over 10 days plus logo in print media daily in two papers in two cities
  Other Names: health promotion; burn prevention

SUMMARY:
The aim of this study was to evaluate the effectiveness of a targeted burn prevention message on burn safety knowledge and behavior.

DETAILED DESCRIPTION:
Flammable liquid burns comprise 23% of admissions to our burn center. This was a project to test the uptake of the message "Don't be a Flaming Fool" delivered via multi-media campaign.

ELIGIBILITY:
Inclusion Criteria:

* male 16 years of age or older

Exclusion criteria

* males less than 16 years of age
* females

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1637 (Actual)
Dates: Start 2010-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Changes in burn safety knowledge at 3 months | Pre intervention, 3 months post intervention
  The changes in knowledge regarding the dangers of using petrol or gasoline before and after a media campaign
Changes in burn safety knowledge at 12 months | pre-intervention and 12 months post-interevention
  The changes in knowledge regarding the dangers of using petrol or gasoline before and after a media campaign

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Muller, FRACS, Principal Investigator — The University of Queensland
Locations (1):
- Royal Brisbane and Women's Hospital, Brisbane, Queensland, Australia